CLINICAL TRIAL: NCT03231566
Title: A Randomized Clinical Trial of Preoperative Pain Neuroscience Education for Total Knee Arthroplasty
Brief Title: Pain Neuroscience Education in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 710848-3
Record Dates: First submitted 2017-07-13; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Total Knee Replacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome measures were mailed by patients in prepaid envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual education control group (CG) (Active Comparator): The CG received the traditional hospital preoperative program, which was consistent with current preoperative TKA protocols. The CG received education covering anatomy of the knee joint, information about the joint replacement surgery, what to expect when they were admitted for surgery, what to expect immediately after surgery, pain medications, postoperative rehabilitation/physical therapy, etc. The CG received a hospital-based booklet with this information.
  Interventions: Behavioral: Pain Neuroscience Education
- Experimental group (EG) (Experimental): The EG underwent an additional 30-minute group PNE program, followed by the usual preoperative education program from the hospital. The PNE program used in this TKA study was an adaptation of the PNE program developed for LS. The educational program was designed to be delivered by a physical therapist in a group session to patients prior to their TKA.
  Interventions: Behavioral: Pain Neuroscience Education

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — See arm/group description

SUMMARY:
To determine if education about pain given prior to Knee Arthroplasty will result in better outcomes following surgery

DETAILED DESCRIPTION:
To determine if a preoperative pain neuroscience education (PNE) program would result in superior outcomes compared to usual preoperative education for total knee arthroplasty (TKA). Patients will receive traditional hospital preoperative TKA program (usual care group) or receive the same program plus an additional 30-minute PNE program (experimental group). Pre and post measurements at 1, 3 and 6 months for pain, function, fear of movement and pain catastrophization. We will also compare opioid usage, healthcare expenses and patient satisfaction between groups.

ELIGIBILITY:
Inclusion Criteria:

* be scheduled to have a TKA and their standard preoperative TKA education program, indicate their willingness to participate in the study, ability to read and understand English, as the study included the use of an educational booklet, and be able and willing to complete outcome data for 6 months after TKA

Exclusion Criteria:

* Because all potential participants for this study had been screened and cleared for their orthopedic surgery, the only exclusion criterion was an unwillingness to participate in the study and having had a previous TKA or scheduled for a bilateral TKA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Pain | Change from Baseline to 1 month, 3 months and 6 months post-surgery
  Numeric Pain Rating Scale
Function | Change from Baseline to 1 month, 3 months and 6 months post-surgery
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Pain Catastrophization | Change from Baseline to 1 month, 3 months and 6 months post-surgery
  Pain Catastrophization Scale
Fear of movement | Change from Baseline to 1 month, 3 months and 6 months post-surgery
  Tampa Scale of Kinesiophobia

SECONDARY OUTCOMES:
Opioid Use | Change at 1 month
  Oral Morphine Dose Equivalents
Healthcare Expenses | Change from Baseline to 1 month, 3 months and 6 months post-surgery
  Costs associated with healthcare utilization
Patient Satisfaction | Change at 1 month, 3 months and 6 months post-surgery
  Likert questions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No